CLINICAL TRIAL: NCT04353115
Title: Usability of a Serious Game to Rehabilitate Gaze Stability in Children with Vestibular Deficit: "Kids Gaze Rehabilitation"
Brief Title: A Serious Game to Rehabilitate Gaze Stability in Children with Vestibular Deficit
Acronym: KG-REHAB
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0692
Record Dates: First submitted 2020-03-02; First posted 2020-04-20 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Vestibular Disorder
Keywords: Vestibular Disorder; serious game; vestibular rehabilitation
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Training with Serious Game: Trained group, 5 weeks training with the serious game; patients have a vestibular impairment.
  Interventions: Device: Training with Serious game

INTERVENTIONS:
Device: Training with Serious game — training the gaze stability with a serious game, 20 minutes a day, 2 days a week for 5 weeks in the presence of a doctor or physiotherapist, at the hospital to avoid addiction at home.

SUMMARY:
Since the early 2000s, vestibular rehabilitation has been proposed as a therapeutic tool to improve the balancing function and the various motor skills in children, in particular in children with hearing loss suffering from concomitant vestibular deficit. It has been demonstrated in adults with vestibular deficit that the fact of adding to the classic exercises on the control of balance per se and habituation, specific exercises of adaptation and substitution of the vestibulo-ocular reflex brought therapeutic benefit. These exercises, which are started in the presence of the physiotherapist and then continued by the patient himself at his home, aim to improve the stabilization of the gaze during head movements. In pediatrics, however, performing them is more difficult than conventional exercises, since their immediate interest is not well understood by the child, who may be reluctant to perform them. The present project aims to enrich the therapeutic offer by a pediatric rehabilitation method of eye stabilization sufficiently playful to win adherence to treatment, including in the absence of the physiotherapist when the child is at home.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a vestibular disorder by the batteries of tests used in clinical routine.
* Supported by the multidisciplinary team of the Audiology and Otoneurological Exploration Department at the HFME
* Patient or parents able to understand the ins and outs of the study
* No opposition from children and parents

Exclusion Criteria:

* Associated visual sensorineural deficit
* Orthopedic or muscular disorder in the cervical spine

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with vestibular disorde
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Numbers of patients able to use the serious game without side effects | Week 5
  the purpose is to defined the proportion of patients able to use the serious game without side effects for 20 minutes a day, 2 days a week for 5 weeks in the presence of a doctor or physiotherapist at the hospital in addition to the usual rehabilitation.

SECONDARY OUTCOMES:
side effects after the 5 weeks of intervention | Week 5
  The side effects collected after the 5 weeks of intervention or at the end of the intervention if it is interrupted before the end are:
  Intolerance to the screen sickness technique, motion sickness type (dizziness, headache, nausea, vomiting, eyestrain, visual disturbances, inability to stand after a session) By means of an adapted questionnaire SSQ (Child Simulator Sickness Questionnaire), adapted and translated into French.
  Values from 0 to 70 : 70 means that childs feel sick
Patient satisfaction | week 5
  Description: will be defined using a Likert scale of faces after each session (5 questions, from 1 to 5 points). 1 being not at all satisfied with the game and 5 being completely satisfied with the game after each session. Suggestions for modifying the game will also be collected
Satisfaction of the patient's parents | Week 5
  Satisfaction of the patient's parents will be defined using a Likert scale of 5 questions out of 5 points, 1 being not at all satisfied with the game and 5 being completely satisfied with the game after each session. Game modification suggestions will also collected
Alouette test | Week 5
  The Alouette test which assesses the fluency in reading questionnaires. The interest of the serious game at the end of the 5 weeks will be evaluated using the comparison between the initial and 5 week evaluation.
Posturo-motor control | Week 5
  The Posturo-motor control with the movement evaluation battery in children M-ABC 2.
  The interest of the serious game at the end of the 5 weeks will be evaluated using the comparison between the initial and 5 week evaluation.
Visual acuity | Week 5
  The interest of the serious game at the end of the 5 weeks will be evaluated using the comparison between the initial and 5 week evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Pr THAI VAN, Bron, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ortega Solis J, Reynard P, Spruyt K, Becaud C, Ionescu E, Thai-Van H. Developing a serious game for gaze stability rehabilitation in children with vestibular hypofunction. J Neuroeng Rehabil. 2023 Sep 26;20(1):128. doi: 10.1186/s12984-023-01249-x. PMID 37752531